CLINICAL TRIAL: NCT06699238
Title: Is There an Anti-inflammatory Effect of Aerobic Exercises on Axial Spondyloarthropathy Patients?: Prospective Randomised Controlled Trial
Brief Title: Effect of Aerobic Exercises on Axial Spondyloarthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeşim Ozge Gunduz Gul (Other Government)
Collaborators: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Yeşim Ozge Gunduz Gul, Resident, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraEtlik-FTR-YOGG-01
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Axial Spondyloarthritis (AxSpA); Aerobic Exercise; Disease Activity
Keywords: axial spondyloarthritis; aerobic exercises; cytokines; acute phase biomarkers; non pharmacological intervention
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups, one group was provided home exercise program and one group run on the treadmill in addition to their home exercise program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Exercise Group (Active Comparator): The home exercise group performed only standard conventional exercises for 12 weeks, 3 days a week, once a day for 30 min, including cervical, thoracic, and lumbar spine flexibility, shoulder muscles, hip flexors, hamstring and quadriceps muscle stretching, spinal flexor stretching, and extensor strengthening and breathing exercises program was shown by the same physician. Patient compliance with the exercise program was monitored weekly using telemedicine.
  Interventions: Other: Home Exercise
- Aerobic Exercise Group (Experimental): The aerobic exercise group performed the following training: warm-up for 5 min, walking for 20 min at an intensity that would use 60-70% of the HR reserve, and cool down for 5 min. Additionally, they performed standard conventional exercises at home for 12 weeks, 3 days a week, once a day for 30 min, including cervical, thoracic, and lumbar spine flexibility, shoulder muscles, hip flexors, hamstring and quadriceps muscle stretching, spinal flexor stretching, and extensor strengthening and breathing exercises program was shown by the same physician. The aerobic exercise group performed on a treadmill under the supervision of a physician.
  Interventions: Other: Home Exercise; Other: Aerobic exercise

INTERVENTIONS:
Other: Home Exercise — Standard conventional exercise for 12 weeks, 3 days a week, once a day for 30 min, including cervical, thoracic, and lumbar spine flexibility, shoulder muscles, hip flexors, hamstring and quadriceps muscle stretching, spinal flexor stretching, and extensor strengthening and breathing exercises program was shown by the same physician. Patient compliance with the exercise program was monitored weekly using telemedicine.
  Other Names: Conventional Exercise
Other: Aerobic exercise — The aerobic exercise group performed the following training: warm-up for 5 min, walking for 20 min at an intensity that would use 60-70% of the HR reserve, and cool down for 5 min. Additionally, they performed standard conventional exercises at home for 12 weeks, 3 days a week, once a day for 30 min, including cervical, thoracic, and lumbar spine flexibility, shoulder muscles, hip flexors, hamstring and quadriceps muscle stretching, spinal flexor stretching, and extensor strengthening and breathing exercises program was shown by the same physician. Patient compliance with the exercise program was monitored weekly using telemedicine.The aerobic exercise group performed on a treadmill under the supervision of a physician.
  Arms: Aerobic Exercise Group

SUMMARY:
This study aimed to examine whether aerobic exercises, in addition to home exercises, have anti-inflammatory effects, which are evaluated by disease activity, acute phase reactants, and cytokine levels in axial spondyloarthropathy

DETAILED DESCRIPTION:
Spondyloarthropathies (SpAs) are a group of chronic, inflammatory, and multisystemic diseases with common genetic, epidemiological, and clinical features. These diseases primarily involve the axial skeleton.

The pathogenesis of SpA is multiple factors. The disease-specific inflammatory response, with the contribution of environmental factors based on genetic predisposition, is responsible for the pathogenesis of the disease.1 The main cytokines thought to be involved in the pathogenesis of axSpa are tumor necrosis factor-alpha (TNF-α), interleukin-17 (IL-17), IL-23, IL-22, IL-6, IL-7, interferon-gamma (IFN-γ), IL-12, and IL-26.

There is no definitive marker associated with disease activity. Studies on cytokine levels and disease activity have shown that TNF-α, IL-6, IL-17, IL-23, and IFN-γ levels may be associated with disease activity in AS patients.4-9 Nonpharmacological and pharmacological methods are used together for the treatment of SpA. Non-pharmacological methods include patient education, smoking cessation, regular exercise, and physiotherapy practices.

Aims of exercise therapy are to improve or preserve range of motion, flexibility, balance and to improve muscle strength and aerobic capacity. Posture, stretching, breathing, strengthening, and aerobic exercises are the most recommended in treating AS.

Exercise therapy is described as the cornerstone treatment of axSpA by the European Alliance of Associations for Rheumatology (EULAR). Although patient compliance with exercise therapy is not easy, the advantages of exercise are that it is cheap, low-risk, and easy to apply compared to pharmacological treatments.

The anti-inflammatory effects of exercise have recently been discussed. Few studies have investigated the anti-inflammatory effects of exercise in patients with AS. While some of these studies showed significant improvement in disease activity, functional status, flexibility, and CRP with aerobic exercise in patients with AS, some did not. Although a few studies have shown a significant decrease in TNF-α levels in AS patients with non-aerobic exercise programs, no study has examined the changes in TNF-α and IL-17 levels with aerobic exercise treatment.

The primary aim of our study was to examine whether aerobic exercise, in addition to the home exercise program, has an anti-inflammatory effect in patients with axSpA, as evaluated by disease activity, acute phase reactants, and cytokine levels. Our secondary aim was to determine whether aerobic exercise, in addition to home exercise, has a positive effect on functional status, functional exercise capacity, quality of life, NSAID consumption, chest expansion, and spinal mobility.

ELIGIBILITY:
Inclusion Criteria:

* AxSpA diagnosis according to the ASAS classification criteria
* Voluntary participation in the study
* Age 20-65 ages
* Regular use of disease-modifying anti-rheumatic drugs at a stable dosage for at least 3 months
* Regular use of NSAID at a stable dosage for at least 4 weeks
* Presence of low disease activity (1.3 ≤ ASDAS-CRP< 2.1)
* Having a phone number that can be used to communicate with oneself or a family member
* At least a primary school graduate.

Exclusion Criteria:

* Presence of active peripheral joint involvement
* Having used a biological agent at any time before
* Exercising regularly for the previous 6 months
* The presence of cardiovascular, orthopedic, and neurological problems that may prevent exercise (unstable angina, uncontrolled sinus tachycardia, presence of severe aortic stenosis, uncontrolled atrial or ventricular arrhythmia, 3rd degree atrioventricular block, fracture, prosthesis, neuropathy, myopathy)
* Any other respiratory or neuromuscular disease that affects the respiratory muscles
* Presence of malignancy
* Presence of pregnancy
* Having undergone any surgery in the previous 6 months,
* Presence of severe psychiatric illness
* Findings related to infection during interrogation
* Having an infection in the last 3 months
* Communication problems
* Having known diabetes mellitus
* The presence of severe comorbidity that may affect the kidneys and livers
* Inability to participate in at least 75% of the exercises
* Having left study voluntarily
* Presence of any new symptoms or findings that develop during exercise or evaluations, and may interfere with exercise.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
ASDAS-CRP | 12 weeks
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is an index to assess disease activity in Ankylosing Spondylitis (AS).
  The prefered score uses CRP.
  ASDAS-CRP = 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1)
  Back pain, patient global assessment, duration of morning stiffness and peripheral pain/swelling are all assessed on a numerical rating scale (from 0 to 10).
  The 3 cut-offs selected to separate these states were: <1.3 between "inactive disease" and "moderate disease activity", <2.1 between "moderate disease activity" and "high disease activity", and >3.5 between "high disease activity" and "very high disease activity".
  Cut-offs for improvement scores were: a change ≥1.1 units for "clinically important improvement"
Tumor necrosis factor-alpha (TNF-α) | 12 weeks
  TNF-α is a chemical messenger produced by the immune system that induces inflammation. Its relation with axial spondyloarthropathy's disease activity is uncertain but inhibition of TNF-α is one of the targets of current therapies. There were no cut-off measures for TNF-α on axial spondyloarthropathy patients.
Interleukin-17 (IL-17) | 12 weeks
  IL-17 is a pro-inflammatory cystine knot cytokines. They are produced by a group of T helper cell known as T helper 17 cell in response to their stimulation with IL-23. Its relation with axial spondyloarthropathy's disease activity is uncertain but inhibition of IL-17 is one of the targets of current therapies. There were no cut-off measures for IL-17 on axial spondyloarthropathy patients.
C-reactive protein (CRP) | 12 weeks
  CRP is an annular (ring-shaped) pentameric protein found in blood plasma, whose circulating concentrations rise in response to inflammation. It is an acute-phase protein of hepatic origin that increases following interleukin-6 secretion by macrophages and T cells. On axial spondyloarthropathy patients it may be elevated but in some patients there could be no elevation of CRP. Also it is necessary for ASDAS-CRP calculation.
Erythrocyte Sedimentation Rate (ESR) | 12 weeks
  Erythrocyte Sedimentation Rate (ESR) is the rate at which red blood cells in anticoagulated whole blood descend in a standardized tube over a period of one hour. On axial spondyloarthropathy patients it may be elevated but in some patients there could be no elevation of ESR. Also it is necessary for disease activity calculation (ASDAS-ESR).

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | 12 weeks
  The visual analogue scale (VAS) is a psychometric response scale that can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. We use the 0-10 cm VAS to measure patients' pain severity. We used 0 as no pain and 10 as unbearable pain.
The Bath Ankylosing Spondylitis Functional Index (BASFI) | 12 weeks
  The Bath Ankylosing Spondylitis Functional Index was named for the location of the institution (Bath, England) where authors A. Calin and co-workers developed this validated index to determine the degree of functional limitation in patients with the inflammatory autoimmune disease Ankylosing Spondylitis (AS). we used BASFI for the patients' functional assessment. BASFI measured by answering a questionaire which has 10 questions about activities of daily life, bending, lie down, position changes, climbing stairs, standing abilities. Then gathered points divided by 10. High scores represents low functional state.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 12 weeks
  BASMI used for all the patients who are attended to our study to assessment of the spinal mobility. BASMI has 3 point scale. BASMI is the most applicated and effective method to assessment of axial mobility. It has five different clinical measurements which are cervical rotation, tragus wall distance, lumbar flexion, trunk lateral flexion, and intermalleolar distance. High scores are associated with poor spinal mobility
Chest expansion measurement | 12 weeks
  Chest expansion is based on the difference between the chest circumference measurement after a deep inspiration at the level of the 4th intercostal space and the chest circumference measurement after a forced expiration. The normal value of chest expansion may vary depending on age and gender. It is expected to be at least 5 cm in young healthy individuals.
6 minute walk test (6 MWT) | 12 weeks
  6 MWT was used to evaluate the functional exercise capacity of the patients participating in the study. While doing 6 MWT, the patients is asked to go as fast as they can between the marked points on at least 30 meters of flat ground, but not to run. Standard commands are used during the test. The total walking distance is recorded for 6 minutes. An increase of 30 meters in 6 MWT is thought to indicate clinical improvement.
Ankylosing Spondylitis Quality of Life (ASQoL) | 12 weeks
  The ASQoL scale was used in the evaluation of the patients participating in the study. This scale consists of 18 questions that can be answered "yes" or "no". 1 point is given for a "yes" answer and 0 point is given for a "no" answer. At the end of the test, all scores are added up. Numerically high results indicate a low quality of life.
Weekly NSAID receive | 12 weeks
  Weekly NSAID receive has obtained by telemedicine both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ajda Bal, MD, Professor, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital Physical Medicine and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No